CLINICAL TRIAL: NCT04528745
Title: The Relationship Between Fat Free Mass and Toxicity of Cytostatics in Cancer Patients
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Jens Rikardt Andersen, Associate Professor, University of Copenhagen
Other Study IDs: H-20000245
Record Dates: First submitted 2020-04-28; First posted 2020-08-27 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Pancreas Cancer; Colorectal Cancer
Keywords: cancer; chemotherapy; toxicity; lean body mass; cytostatics; fat free mass; dose-limiting toxicity; adverse events; adult; quality of life; nutrition
MeSH Terms: conditions — Pancreatic Neoplasms; Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cancer receiving cytostatic treatment: Consecutive patients referred for cytostatic treatment or in treatment with cytostatic agents for colorectal or pancreatic cancer
  Interventions: Diagnostic Test: Bio Impedance Spectroscopy (BIS)

INTERVENTIONS:
Diagnostic Test: Bio Impedance Spectroscopy (BIS) — Determination of fat free mass by BIS

SUMMARY:
An observational study of the relationship between fat free mass and toxicity of cytostatics in cancer patients, at the department of Clinical Oncology at Zealand University Hospital, Roskilde, Denmark. Fat free mass will be measured by bio impedance spectroscopy and data on toxicity will be obtained from medical records and interviews/questionnaires with the patients.

DETAILED DESCRIPTION:
With a prospective observational design, this study will examine whether there is a correlation between the total dose of cytostatics per measured fat-free mass (FFM) (mg cytostatic agent/kg FFM) and toxicity of cytostatics among cancer patients. The study will include patients with a primary diagnosis of any stage colorectal or pancreatic cancer.

The hypothesis is, that a higher total dose of cytostatics per FFM will correlate to more frequent and/or more severe toxicity than a lower total dose. In extension to this, we hypothesize that a loss of FFM during treatment, and thereby an increased total dose of cytostatics per FFM, will lead to more frequent and severe toxicity.

Recruitment and data collection will take place at the department of Clinical Oncology at Zealand University Hospital, Roskilde over about a five month period. Each patient will be included for two-four cycles of cytostatic treatment. FFM will be measured by bio impedance spectroscopy as close to the first day of each cycle of cytostatic treatment as possible. Information about toxicity will be obtained from patient records and through interviews with the patients. Interviews will be conducted at day 5 (4-6) of each cycle and at the end of each cycle. The interviews include questionnaires about specific toxicities, using National Cancer Institute (NCI) Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE), and overall health and quality of life, and 24-hour recall of dietary intake and questions about physical activity level.

In short, relevant outcomes are change in FFM, hematology, grade 3/4 hematological toxicity as defined by NCI CTCAE, dose-limiting toxicity, hospitalization, patient-reported adverse events, overall health and quality of life, and nutritional intake.

ELIGIBILITY:
Inclusion Criteria:

* Authorized individuals
* Understands, speaks and reads Danish
* Patients referred for or who receives cytostatic treatment, and have a primary diagnosis of colorectal- or pancreatic cancer (diagnoses classified by International Classification of Diseases-10 as C18-21 and C25)
* Have the possibility of contact by telephone

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Dementia
* Contraindications for BIS measuring (pacemaker)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at the department of Clinical Oncology at Zealand University Hospital, Roskilde, Denmark, who fulfills all inclusion criteria and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Change in fat free mass between cycles of cytostatic treatment (each cycle lasts for 14, 21 or 28 days, depending on the type of regime) | During and between two-four cycles, depending on regime (each cycle is 14, 21 or 28 days, depending on the regime)
  Changes in fat free mass, measured at baseline and the beginning of each cycle, between cycles of cytostatic treatment, and correlation with dose of cytostatic agent (mg) pr. fat free mass (kg)
Leucocyte count (per cycle - see outcome 1) | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between change i absolute and relative leucocyte count from baseline, and total dose of cytostatic agent (mg) pr. fat free mass (kg)
Thrombocyte count (per cycle - see outcome 1) | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between change i absolute and relative thrombocyte count from baseline, and total dose of cytostatic agent (mg) pr. fat free mass (kg)
Mmol of haemoglobin/L (per cycle - see outcome 1) | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between change i absolute and relative mmol of haemoglobin/L from baseline, and total dose of cytostatic agent (mg) pr. fat free mass (kg)
Neutropenia | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between incidence of absolute neutrophilic granulocyte count <1.0 - 0.5 x 10e9/L and total dose of cytostatic agent (mg) pr. fat free mass (kg)
Febrile neutropenia | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between incidence of absolute neutrophilic granulocyte count <1.0 x 10e9/L, with a single temperature of >38.3 degrees C or a temperature of >= 38 degrees C lasting for more than one hour, and total dose of cytostatic agent (mg) pr. fat free mass (kg)
Anemia | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between incidence of haemoglobin <4,9 mmol/L(; transfusion indicated) and total dose of cytostatic agent (mg) pr. fat free mass (kg)
Thrombocytopenia | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between incidence of absolute thrombocyte count <50.0 - 25.0 x 10e9 /L and total dose of cytostatic agent (mg) pr. fat free mass (kg)

SECONDARY OUTCOMES:
Dose-limiting toxicity (DLT) | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between DLT and total dose of cytostatic agent (mg) pr. fat free mass (kg).
  DLT is defined as toxicity leading to one or more of the following: Dose reduction of one or more cytostatic agent(s) (recorded as mg and %). Postponement of cytostatic therapy (recorded as number of days). Discontinuation of cytostatic therapy before scheduled.
  Causes of DLT (that are registered in patients records) are classified in one or more of the following categories: Infection, organ impact, myelosuppression, gastrointestinal discomfort, neuropathy or other toxicity (which one is recorded).
Hospitalization | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Hospitalization note in patient record. Correlation between incidence and number of days of hospitalization and total dose of cytostatic agent (mg) pr. fat free mass (kg).

OTHER OUTCOMES:
Overall health | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between overall health, and change therein, the first 5 (4-6) days of a cycle or the last week of a cycle, evaluated on a 7-point scale, and total dose of cytostatic agent (mg) pr. fat free mass (kg).
Overall quality of life | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between overall quality of life, and change therein, the first 5 (4-6) days of a cycle or the last week of a cycle, evaluated on a 7-point scale, and total dose of cytostatic agent (mg) pr. fat free mass (kg).
Energy intake (per cycle - see outcome 1) | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between relative fulfilment of energy requirement, and change therein, on day 5 (4-6) of a cycle or the last day of a cycle, and total dose of cytostatic agent (mg) pr. fat free mass (kg), and change in fat free mass (kg). Energy requirement is estimated by Harris-Benedict formula, including among other assessment of physical activity level. Energy intake is assessed by 24-hour recall of nutrition intake.
Protein intake (per cycle - see outcome 1) | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between relative fulfilment of protein requirement, and change therein, on day 5 (4-6) of a cycle or the last day of a cycle, and total dose of cytostatic agent (mg) pr. fat free mass (kg), and change in fat free mass (kg). Protein requirement is estimated from the Danish Health Authority´s recommendation for adult patients. Protein intake is assessed by 24-hour recall of nutrition intake.
Weight change (per cycle - see outcome 1) | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between relative and absolute weight change, measured at the beginning of each cycle, and total dose of cytostatic agent (mg) pr. fat free mass (kg), and change in fat free mass (kg).
Difficulty swallowing | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between patient reported severity and interference with daily activities of difficulty swallowing on a 5-point scale, and change therein, the last week of a cycle, and total dose of cytostatic agent (mg) pr. fat free mass (kg).
Mouth/throat sores | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between patient reported severity and interference with daily activities of mouth/throat sores on a 5-point scale, and change therein, the last week of a cycle, and total dose of cytostatic agent (mg) pr. fat free mass (kg).
Taste changes | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between patient reported severity of taste changes on a 5-point scale, and change therein, the last week of a cycle, and total dose of cytostatic agent (mg) pr. fat free mass (kg).
Decreased appetite | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between patient reported severity and interference with daily activities of decreased appetite on a 5-point scale, and change therein, the first 5 (4-6) days of a cycle or the last week of a cycle, and total dose of cytostatic agent (mg) pr. fat free mass (kg).
Nausea | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between patient reported frequency and severity of nausea on a 5-point scale, and change therein, the first 5 (4-6) days of a cycle or the last week of a cycle, and total dose of cytostatic agent (mg) pr. fat free mass (kg).
Vomiting | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between patient reported frequency and severity of vomiting on a 5-point scale, and change therein, the first 5 (4-6) days of a cycle or the last week of a cycle, and total dose of cytostatic agent (mg) pr. fat free mass (kg).
Constipation | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between patient reported severity of constipation on a 5-point scale, and change therein, the last week of a cycle, and total dose of cytostatic agent (mg) pr. fat free mass (kg).
Diarrhea | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between patient reported frequency of diarrhea on a 5-point scale, and change therein, the first 5 (4-6) days of a cycle or the last week of a cycle, and total dose of cytostatic agent (mg) pr. fat free mass (kg).
Shortness of breath | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between patient reported severity and interference with daily activities of shortness of breath on a 5-point scale, and change therein, the last week of a cycle, and total dose of cytostatic agent (mg) pr. fat free mass (kg).
Rash | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between patient reported incidence of rash (yes/no), and change therein, of the last week of a cycle, and total dose of cytostatic agent (mg) pr. fat free mass (kg).
Hair loss | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between patient reported degree of hair loss on a 5-point scale, and change therein, the last week of a cycle, and total dose of cytostatic agent (mg) pr. fat free mass (kg).
Hand-foot syndrome | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between patient reported severity of hand-foot syndrome on a 5-point scale, and change therein, the last week of a cycle, and total dose of cytostatic agent (mg) pr. fat free mass (kg).
Numbness & tingling | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between patient reported severity and interference with daily activities of numbness and tingling on a 5-point scale, and change therein, the first 5 (4-6) days of a cycle or the last week of a cycle, and total dose of cytostatic agent (mg) pr. fat free mass (kg).
General pain | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between patient reported frequency, severity and interference with daily activities of general pain on a 5-point scale, and change therein, the first 5 (4-6) days of a cycle or the last week of a cycle, and total dose of cytostatic agent (mg) pr. fat free mass (kg).
Fatigue | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between patient reported severity and interference with daily activities of fatigue on a 5-point scale, and change therein, the last week of a cycle, and total dose of cytostatic agent (mg) pr. fat free mass (kg).
Nosebleed | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between patient reported frequency and severity of nosebleed on a 5-point scale, and change therein, the last week of a cycle, and total dose of cytostatic agent (mg) pr. fat free mass (kg).
Other adverse event(s) added by patient | During two-four cycles, depending on regime (about eight-nine weeks), and within each cycle (each cycle is 14, 21 or 28 days)
  Correlation between patient reported severity of adverse event(s) on a 5-point scale, and change therein, the first 5 (4-6) days of a cycle or the last week of a cycle, and total dose of cytostatic agent (mg) pr. fat free mass (kg).

CONTACTS AND LOCATIONS:
Overall Officials: Jens R Andersen, Principal Investigator — University of Copenhagen
Locations (1):
- Zealand University Hospital, Roskilde, Denmark